CLINICAL TRIAL: NCT04454398
Title: A Randomized, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics and Efficacy of a Single Dose of STI-1499 (COVI-GUARD™) in Hospitalized Patients With Moderate COVID-19
Brief Title: Study to Evaluate STI-1499 (COVI-GUARD) in Patients With Moderate COVID-19
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GRD-COV-101
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — STI-2020; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- COVI-GUARD (Experimental): COVI-GUARD (STI-1499) administered via a single IV push injection at a dose of 10 mg, 30 mg, 100 mg, or 200 mg, in addition to standard of care
  Interventions: Biological: COVI-GUARD; Other: Standard of Care
- Placebo (Placebo Comparator): Placebo administered via a single IV push injection, in addition to standard of care
  Interventions: Other: Standard of Care; Drug: Placebo

INTERVENTIONS:
Biological: COVI-GUARD — COVI-GUARD (STI-1499) is a monoclonal antibody which targets the COVID-19 spike protein
  Other Names: STI-1499
  Arms: COVI-GUARD
Other: Standard of Care — Standard of Care as determined by the Investigator
Drug: Placebo — Diluent
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled study to evaluate the safety, pharmacokinetics and efficacy of a single dose of STI-1499 (COVI-GUARD™) in hospitalized patients with moderate COVID-19

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled study to evaluate the safety, pharmacokinetics and efficacy of a single dose of STI-1499 (COVI-GUARD™), a COVID-19 targeting monoclonal antibody, in hospitalized patients with moderate COVID-19. Four dose levels will be tested: 10 mg, 30 mg, 100 mg, and 200 mg.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of moderate COVID-19, diagnosed standard RT-PCR assay or equivalent testing
* Willing and able to comply with study procedures and follow-up visits
* Subject or family member/caregiver must have provided written informed consent which includes signing the institutional review board approved consent form prior to participating in any study related activity. However, if obtaining written informed consent is not possible, other procedures as provided in the March 27th, 2020 FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Pandemic, Question 10, may be used.

Exclusion Criteria:

* Clinical signs indicative of severe COVID-19
* Rapidly progressive COVID-19 which is likely to progress to "severe" within 24 hours
* Documented infection other than COVID-19
* Any medical condition that, in the Investigator's opinion, could adversely impact safety
* Pregnant or lactating women
* Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, monoclonal antibodies (mAbs) against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit. Note: Participants who have been prescribed hydroxychloroquine or chloroquine with or without azithromycin or other approved products for the off-label treatment of COVID-19 prior to study enrollment may be included and may continue to receive these agents so long as the dose remains stable. Additionally, any approved or authorized treatment (e.g., remdesivir, dexamethasone or treatments approved under an Emergency Use Authorization) is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (safety) | Randomization through study completion through Day 60
  Types, frequencies, and severities of adverse events and their relationships to COVI-GUARD
Incidence of treatment-emergent adverse events (safety) | Randomization through study completion through Day 60
  Types, frequencies, and severities of treatment-emergent adverse events and their relationships to COVI-GUARD
Incidence of serious adverse events (safety) | Randomization through study completion through Day 60
  Types, frequencies, and severities of serious adverse events and their relationships to COVI-GUARD
All-cause mortality at 29 and 60 days | Randomization through Day 29 and Day 60
  All-cause mortality at 29 and 60 days
Incidence of dose-limiting toxicities (safety) | Randomization through study completion through Day 60
  Dose-limiting toxicities, particularly presence of acute or delayed hypersensitivity reactions
Incidence of laboratory abnormalities (safety) | Randomization through study completion through Day 60
  Clinically meaningful laboratory abnormalities
SARS-CoV-2 viral load as assessed using various sample types | Randomization through study completion through Day 60
  Plasma samples and salivary samples are taken to correlate viral load with nasopharyngeal testing at various timepoints; stool or rectal swab samples are taken if possible for additional virologic assessments
Time to hospitalization, treatment, ICU admission, and discharge from ICU and/or hospital | Randomization up to study completion through Day 60
  Time from onset of COVID-19 symptoms to hospitalization and to treatment on Day 1, and if applicable, time to ICU admission, discharge from ICU and discharge from hospital
Anti-drug antibodies | Randomization through study completion through Day 60
  Presence and levels of anti-drug antibodies (ADA) directed to COVI-GUARD
Cytokine levels | Randomization through study completion through Day 60
  Levels of cytokines including EGF, IFNγ, IL-1β, IL-6, IL-8, IL-10, and TNFα

SECONDARY OUTCOMES:
AUC of COVI-GUARD (PK) | Randomization through study completion through Day 60
  Area under the serum concentration-time curve (AUC) of COVI-GUARD
Cmax of COVI-GUARD (PK) | Randomization through study completion through Day 60
  Maximum observed serum concentration (Cmax) of COVI-GUARD
t½ of COVI-GUARD (PK) | Randomization through study completion through Day 60
  Apparent serum terminal elimination half life (t½) of COVI-GUARD
Tmax of COVI-GUARD (PK) | Randomization through study completion through Day 60
  Time to Cmax (Tmax) of COVI-GUARD

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343